CLINICAL TRIAL: NCT00766597
Title: Phase I/II Open-Label Study to Evaluate the PK, Safety, Tolerability and Antiviral Activity of Vicriviroc, a Novel CCR5 Antagonist in Combination Regimens in HIV-Infected ART Experienced Children and Adolescents
Brief Title: Safety and Immune Response to Vicriviroc in Combination Regimens in HIV-Infected ART Experienced Children and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1071; 10634 (Registry Identifier: DAIDS ES); IMPAACT P1071
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2015-12

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — vicriviroc

ARMS (1):
- Vicriviroc in tablet form (20/30 mg) or liquid form (1 mg/ml) (Experimental): HIV-1 Infected Antiretroviral Therapy Experienced Participants with CCR5-tropic Virus
  Interventions: Drug: Vicriviroc

INTERVENTIONS:
Drug: Vicriviroc — Administered orally in either tablet or liquid form at a dosage of approximately 0.8/mg/kg every 24 hours, with a ritonavir boosted protease inhibitor containing background regimen

SUMMARY:
Complications with current HIV antiretroviral therapy have left many children and adolescents with limited therapeutic options due to drug resistance. The purpose of this study is to test the effectiveness and safety of Vicriviroc (VCV), an HIV entry inhibitor and CCR5 co-receptor antagonist.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) that includes a protease inhibitor (PI) or a non-nucleoside reverse transcriptase inhibitor (NNRTI) has become the standard treatment of HIV-infected adults and children. When effective, HAART decreases the viral population, increases the body's immune responses, and leads to decreased disease progression and increased survival. However, several factors including poor adherence, drug toxicities, and drug resistance complicate HIV management and allow for children and adolescents to develop resistance to multiple drug classes, leaving them with very limited therapeutic options. Fortunately, drugs with new mechanisms of action, such as HIV entry inhibitors, demonstrate activity even in people with resistance to the currently available reverse transcriptase and protease inhibitors.

The purpose of this study is to test the effectiveness and safety of Vicriviroc (VCV), an HIV entry inhibitor. Vicriviroc targets the CCR5 chemokine receptor, which HIV uses to bind and enter CD4+ cells.

This study is a two-stage, age-stratified, non-comparative study to explore the safety, tolerability, pharmacokinetic profile and antiviral activity of the investigational CCR5 inhibitor Vicriviroc in HIV-infected treatment experienced children and adolescents.

In Step I participants will be screened for the co-receptor CCR5 to assess whether they can enter Step II. Only participants with CCR5-tropic virus are eligible for Step II - the main portion of the study to evaluate the study outcome measures. Those participants who continue to Step II will be assigned to one of four age-stratifies cohorts which will receive varying forms, either liquid or tablet, of Vicriviroc:

Cohort I: 12 years to less than 19 years of age, to receive tablet formulation of VCV

Cohort II: 6 years to less than 12 years of age, to receive tablet formulation of VCV

Cohort III: 6 years to less than 12 years of age, to receive liquid formulation of VCV

Cohort IV: 2 years to less than 6 years of age, to receive liquid formulation of VCV

Dose strengths of 20 mg and 30 mg will be used, or in liquid formulation at a concentration of 1mg/mL.

Step II is composed of Stage I and Stage II. Stage I is a dose ranging study designed to explore how the body responds to different doses of vicriviroc, including safety factors associated with dosage. After optimal dosage information and safety measures have been assessed for the different cohorts in Stage I, Stage II will open. Stage II will evaluate the long term safety, tolerability and effectiveness of vicriviroc.

The study, including Steps I and II will last for approximately 48 weeks. Follow-up for all subjects exposed to vicriviroc will last for 5 years after initial exposure. Visits will be every 3 months for subjects on study provided vicriviroc and every 6 months for subjects who discontinue vicriviroc.

The study was terminated shortly after the initiation, when the drug company decided to discontinue development of the study drug. As of study termination, nine participants had enrolled under Cohort I in Step I, but only 4 participants had CCR5 tropism and received the study medication under Step II. All 4 participants had limited post-baseline data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Treatment experienced subjects: Children or adolescents on an unchanged therapeutic regimen for at least 12 weeks and experiencing virologic failure OR participants on no treatment for 4 weeks or more but with history of virologic failure on a prior therapeutic regimen.
* Likely to have virus that is sensitive to at least one ritonavir boosted protease inhibitor
* HIV viral load greater than or equal to 1,000 copies/ml within 90 days prior to Step I entry
* Able to swallow study medication, in tablets or liquid form specific to age-assigned cohort
* Parent, legal guardian or participant able and willing to provide signed informed consent and to have the participant followed at the clinic site
* Willing to use effective methods of contraception

Inclusion Criteria for Step II (In addition to the inclusion criteria for Step I):

* Participant's plasma HIV tested at Step I must be R5 tropic
* Genotypic sensitivity enabling the participant to take optimized background therapy (OBT) consisting of at least a ritonavir-based protease inhibitor. More information on this criterion can be found in the study protocol.

Exclusion Criteria:

* Presence of any currently active AIDS defining illness or history of malignancy
* History of a seizure disorder that requires current anti-seizure medication for control or at risk for seizures. Those with a history of febrile seizures alone are not excluded.
* Certain abnormal laboratory values. More information on this criterion can be found in the protocol.
* Any vaccinations 14 days prior to Step I, or scheduled to occur within 14 days prior to entry into Step II, and the week 24 and 48 visits in Step II
* Allergy or sensitivity to study drug or its ingredients
* Taking any Step II disallowed medications (see protocol) and unable or unwilling to discontinue them at least one week prior to entering Step II
* Use of NNRTIs other than etravirine 21 days prior to Step II entry
* Pregnancy or breastfeeding. Infants who are receiving breastmilk are allowed to enroll.

Exclusion Criteria for Step II

* All exclusion criteria for Step I
* Participants harboring dual or mixed tropic virus (R5/X4) or X4 virus or non phenotypable virus
* Current or anticipated use of any disallowed medications
* Use of efavirenz, nevirapine, and delavirdine for 21 days prior to Step II entry
* Pregnant within 3 days of Step II entry

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolando M Viani, M.D., M.T.P., Study Chair — University of California; Stephen A Spector, M.D., Study Chair — University of California, San Diego
Locations (9):
- United States (8):
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Chicago Children's CRS, Chicago, Illinois
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Lorenzen T, Stoehr A, Walther I, Plettenberg A. CCR5 antagonists in the treatment of treatment-experienced patients infected with CCR5 tropic HIV-1. Eur J Med Res. 2007 Oct 15;12(9):419-25. PMID 17933723
- [Background] Rusconi S, Scozzafava A, Mastrolorenzo A, Supuran CT. An update in the development of HIV entry inhibitors. Curr Top Med Chem. 2007;7(13):1273-89. doi: 10.2174/156802607781212239. PMID 17627557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine participants were recruited in 9 US sites between Sept 21, 2009 to June 16, 2010 prior to the early study closure on August 10, 2010.
Pre-assignment Details: In Step I, 9 participants under Cohort I were screened for evaluation for co-receptor tropism. Five participants did not have the required tropism and were discontinued from the study. Only 4 participants had the CCR-5-tropic virus tropism, and thus were eligible to go to Step II and were assigned to receive the study drug.
Period: Overall Study
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Started | 9 (Screened participants who were evaluated for co-receptor tropism)
With CCR5-tropic Virus | 4 (Evaluable participants, received the study drug)
Without CCR5-tropic Virus | 5 (Not evaluable participants, did not receive the study drug)
Completed Week 24 | 1 (Week 24 is the first primary time point of analysis)
Completed Week 48 | 0 (Week 48 is the second primary time point of analysis)
Completed | 0 (Treatment duration is 48 weeks plus 5 years of follow-up)
Not Completed | 9
Not completed — Unexpected closure of study | 4
Not completed — Without CCR5-tropic virus | 5

BASELINE CHARACTERISTICS:
Population: The HIV-1 infected antiretroviral therapy experienced participants With CCR5-tropic virus who started treatment in Step II
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suspected Adverse Drug Reaction Leading to Treatment Termination
Description: The protocol required reporting of signs and symptoms and laboratory abnormalities of >=Grade 2 and all grades of fever. The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs. Expedited adverse event reporting followed Version 2.0 of the DAIDS Expedited Adverse Event Manual.The attribution of relationship of serious adverse events to study drug for the purposes of employing the start, stop and pause rules is to be determined by the Study Team. Gradation of relationship will use the following terminology: Not related, Probably not related, Possibly related, Probably related or Definitely related.
Time Frame: From study entry to Week 24 or the early study termination whichever occurred earlier
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1mg/ml): HIV-1 Infected Antiretroviral Therapy Experienced Participants with CCR5-tropic virus
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1mg/ml)
Number analyzed (Participants) | 4
participants | 0

2. Primary Outcome: Number of Participants With Adverse Events of Grade 3 or Higher Severity
Description: Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004, Clarification August 2009, which is available on the RCC website at (http://rcc.tech-res.com/). All grade 3 and higher signs, symptoms, and laboratory toxicities were included.
Time Frame: From study entry to Week 24 or the early study termination whichever occurred earlier
Population: The HIV-1 infected antiretroviral therapy experienced participants with CCR-5 tropic virus who started treatment in Step II
Measure: Number; unit: participants
Groups:
- Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1mg/ml): HIV-1 Infected Antiretroviral Therapy Experienced Participants with CCR5-tropic Virus
  Vicriviroc: Administered orally in either tablet or liquid form at a dosage of approximately 0.8/mg/kg every 24 hours, with a ritonavir boosted protease inhibitor containing background regimen
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1mg/ml)
Number analyzed (Participants) | 4
participants | 1

3. Primary Outcome: Number of Participants Who Failed to Meet PK Targets
Description: For Stage I subjects who are enrolled in Step II, the average of the pre-dose and 24 hour post dose sample from the intensive PK evaluations of said subjects will be used as the estimate of Cmin. The whole cohort will fail the PK targets if the population target (median vicriviroc Cmin should be =>200 ng/mL) is not met, and that nearly all of subjects' Cmin failed to be > 100 ng/mL.
Time Frame: At Week 24
Population: The HIV-1 infected antiretroviral therapy experienced participants with CCR-5 tropic virus who started treatment in Step II and who failed the PK targets. Outcome measure not analyzed since the PK targets were for the whole cohort, but the lone cohort opened was not fully enrolled due to early study termination.
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1mg/ml)
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Who Failed to Achieve =>1-log Drop From Baseline in HIV-1 Viral Load and HIV-1 Viral Load of =>400 Copies/mL (Virologic Failures)
Description: Plasma HIV RNA (RNA) concentrations were determined at entry and at regular intervals using the HIV-1 MONITOR Test, version 1.5 (Roche Molecular Diagnostics) or RealTime HIV-1 (Abbott Molecular). The primary definition of virologic success will require subjects to have achieved and maintained 1-log drops from baseline of HIV-1 RNA or HIV-1 RNA <400 copies/mL.
Time Frame: At Baseline, Week 24
Population: HIV-1 infected ART-experienced participants with CCR5-tropic virus who started treatment in Step II and have reached Week 24. Measure was not analyzed since only one participant reached Week 24, no aggregate results were available for posting, and the individual participant-level data were not posted due to being potentially identifiable.
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1mg/ml)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Changes in Co-receptor Tropism From Baseline
Description: Among all patients enrolled in Step I, the prevalence of detectable coreceptor phenotype, R5 tropic, R5/X4 mixed and X4 tropic viruses will be evaluated. The extent to which coreceptor phenotype in Step I is associated with Step I CD4 cell count, HIV RNA, and age will be evaluated. The association of Step I coreceptor phenotype and nadir CD4, HIV subtype, number of ART regimens, and years of ART will be evaluated. At the time of virologic failure, the extent of change from Step I and/or baseline R5 tropic virus to R5/X4 mixed or to X4 tropic virus as detected by the TrofileTM assay will be evaluated.
Time Frame: At Baseline, Week 24
Population: as for outcome 4
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in CD4 Counts
Description: Change in CD4 count from baseline to weeks 24 will be presented both in the aggregate and broken down by age cohort.
Time Frame: At Baseline, Week 24
Population: as for outcome 4
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in CD4 Percent
Description: Change in CD4 percent from baseline to weeks 24 will be presented both in the aggregate and broken down by age cohort.
Time Frame: At Baseline, Week 24
Population: as for outcome 4
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Polymerase Genome and Envelope Sequence
Description: Number of subjects with changes in genotypic and phenotypic drug resistance to the OBT and to vicriviroc (envelope sequence) from baseline to Week 24 and/or virologic failure will be presented both in the aggregate and broken down by age cohort.
Time Frame: At Baseline, Week 24
Population: as for outcome 4
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Plasma HIV RNA PCR
Description: Changes in HIV RNA (copies/mL) from baseline to Week 24 will be presented both in the aggregate and broken down by age cohort.
Time Frame: At Baseline, Week 24
Population: as for outcome 4
Arm/Group | Vicriviroc in Tablet Form (20/30 mg) or Liquid Form (1 mg/ml)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From study entry to the very early study discontinuation
Description: Adverse event summary pertains to the 4 participants accrued into Step I and then into Step II and treated with the study medication.
Groups:
- Vicriviroc in Tablet Form (20/30mg) or Liquid Form (1mg/ml): Drug: Vicriviroc Administered orally in either tablet or liquid form at a dosage of approximately 0.8/mg/kg every 24 hours, with a ritonavir boosted protease inhibitor containing background regimen
Arm/Group | Vicriviroc in Tablet Form (20/30mg) or Liquid Form (1mg/ml)
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vicriviroc in Tablet Form (20/30mg) or Liquid Form (1mg/ml) (N=4)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Eyelid oedema (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Acarodermatitis (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Blood bicarbonate abnormal (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood glucose decreased (Investigations) | 3
Blood glucose increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Genital rash (Reproductive system and breast disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated early with Merck's announcement on July 15, 2010 on the discontinuation of the development of Vicriviroc, with 4 participants given study drug and only 1 participant reached Week 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.